CLINICAL TRIAL: NCT04600089
Title: A Randomized, Double-blind, Placebo-controlled, Study to Identify the Opioid-sparing Effects, and Pain-reduction Potential of Low Dose Ketamine on Patients Undergoing TEVAR Procedures Receiving NCI
Brief Title: Ketamine in Patients Undergoing TEVAR Procedures Receiving NCI
Acronym: 2020Ketamine
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sam Tyagi (Other)
Responsible Party: Sponsor-Investigator, Sam Tyagi, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 60617
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Descending Aortic Dissection; Postoperative Pain; Thoracoabdominal Aortic Aneurysm
Keywords: naloxone; ketamine; aortic repair; spinal cord ischemia
MeSH Terms: conditions — Pain, Postoperative; Aortic Aneurysm, Thoracoabdominal; Spinal Cord Ischemia | interventions — Sodium Chloride; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care (Placebo Comparator): Participants in this group will receive standard of care as well as a saline infusion during the study period.
  Interventions: Drug: Saline
- Sub-Dissociative Ketamine (Experimental): Participants in this group will receive standard of care as well as a continuous ketamine infusion at the induction of anesthesia and for 48 hours postoperatively.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Saline — Saline infusion
  Arms: Standard of Care
Drug: Ketamine — Continuous ketamine infusion at a dose of 0.2 mg/kg/hr, initiated at the induction of anesthesia and continued for 48 hours postoperatively.
  Arms: Sub-Dissociative Ketamine

SUMMARY:
The objective of this study is to identify the opioid-sparing effects, and pain-reduction potential of low dose, sub-dissociative ketamine on patients undergoing thoracic endovascular aortic repair (TEVAR) procedures receiving naloxone continuous infusion (NCI).

DETAILED DESCRIPTION:
Patients undergoing descending aortic repair often experience post-operative pain, and have high post operative opioid requirements. That pain is partially due to the use of naloxone continuous infusion (NCI). NCI is part of a bundled approach used in the first 48 hours post-operatively to prevent spinal cord ischemia, a devastating complication associated with surgical repair of the descending aortic. Data indicate that patients receiving NCI experience elevated post-operative pain scores and increased opioid requirements during the 48-hr post-operative NCI administration, compared to patients not receiving NCI.

Ketamine is an FDA-approved N-methyl D-aspartate (NMDA) antagonist that has been shown to provide adjunctive analgesia and opioid-sparing effects in post-operative surgical patients. At low doses, ketamine provides analgesic benefit without the anesthetic effects seen at higher doses. These doses are commonly referred to sub-dissociative. This study will evaluate whether use of sub dissociative ketamine (SDK) in patients undergoing aortic procedures with the use of NCI will lead to decreased post-operative opioid consumption, and produce improved pain scores in the first 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* willing to give informed consent
* scheduled for elective thoracic aorta repair or thoracoabdominal aortic repair
* requires naloxone continuous infusion for spinal prophylaxis

Exclusion Criteria:

* allergy to ketamine, acetaminophen, or fentanyl
* diagnosis of schizophrenia
* history of hydrocephalus or central nervous system mass
* incarcerated individuals
* pregnant or lactating individuals

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Cumulative Opioid Dose | 48 hours
  Total morphine milligram equivalents (MME) will be assessed every 6 hours for 48 hours.

SECONDARY OUTCOMES:
Change in Pain | 48 hours
  Pain will be assessed using a 10-Point Numerical Pain Scale (as part of standard of care) every hour for the first 24 hours and every two hours for the next 24 hours. Scores range from 0-10; higher scores indicated higher levels of pain.
Number of Patients with Ketamine-Induced Delirium | 48 hours
  Ketamine-induced delirium will be monitored via the Confusion Assessment Method (CAM-ICU) survey every 8 hours for 48 hours. The CAM-ICU assesses four diagnostic features of delirium and the result is a binary (yes or no) determination.
Number of Patients with Uncontrolled Hypertension | 48 hours
  Uncontrolled hypertension is defined as a systolic pressure of 160 mmHg despite 3 intravenous antihypertensive agents.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Rockich, Pharm D, Study Director — University of Kentucky; Samuel Tyagi, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No